CLINICAL TRIAL: NCT03308019
Title: Effectiveness of Scaling and Root Planing With and Without Adjunct Antimicrobial Photodynamic Therapy in the Treatment of Chronic Periodontitis Among Cigarette-smokers and Never-smokers: A Randomized Controlled Clinical Trial
Brief Title: Adjunct Photodynamic Therapy in Chronic Periodontitis Among Cigarette-smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Zohaib Akram, Director, Clinical Research, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FR-17-87
Record Dates: First submitted 2017-10-03; First posted 2017-10-12 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Chronic Periodontitis; Smoking
MeSH Terms: conditions — Chronic Periodontitis; Smoking | interventions — Photochemotherapy; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adjunctive photodynamic therapy (Experimental): This arm will be given scaling and root planing (SRP) with adjunctive photodynamic therapy (aPDT)
  Interventions: Device: Photodynamic therapy; Procedure: Scaling and root planing (SRP)
- Dental scaling (Active Comparator): This arm will be given scaling and root planing (SRP) only
  Interventions: Device: Photodynamic therapy; Procedure: Scaling and root planing (SRP)

INTERVENTIONS:
Device: Photodynamic therapy — In groups 1 and 2, aPDT was performed after SRP. The protocol for aPDT is described elsewhere. Briefly, using a blunt needle, 0.005% of Methylene blue was applied into the periodontal pocket and left in place for 10 seconds. The dye was then irradiated with a diode laser (670 nanometers) at 150 milliwatts. In each dye filled periodontal pocket, laser irradiation was performed for one minute using a flexible tip. In the present study, aPDT was performed once, at baseline, by a trained dentist.
Procedure: Scaling and root planing (SRP) — In both groups, SRP was performed in one session under local anesthesia using handheld Gracey curettes No. 5/6. One trained dental hygienist blinded to the study groups and subgroups made 9 to 10 strokes in a vertical (apico-coronal) direction and the inclination between scaler tips and roots was maintained as zero. When the curved explorer indicated a smooth and hard dental surface, SRP was judged as completed. In all individuals, SRP was done in one session without any assigned time limit for completion.

SUMMARY:
This study evaluates the efficacy of scaling and root planing with and without adjunct antimicrobial photodynamic therapy (aPDT) in the treatment of chronic periodontitis (CP) among cigarette-smokers and never-smokers.

DETAILED DESCRIPTION:
The following inclusion criteria were entailed: (a) Self-reported habitual cigarette-smokers; (b) self-reported never-smokers; (c) patients with CP (presence of at least 30% sites with ≥ 3 mm of CAL and PD ≥ 3 mm 18, 19 ). The exclusion criteria were as follows: (a) patients with systemic diseases such as acquired immune deficiency syndrome/HIV and diabetes mellitus; (b) habitual smokeless tobacco product and alcohol users; (c) third molars and fractured teeth with embedded root remnants and edentulous individuals; (d) patients with misaligned teeth; and (e) patients that reported to have used antibiotics, non-steroidal anti-inflammatory drugs and/or steroids within the past 90 days.

Demographic information was collected using a questionnaire. Cigarette-smokers (group-1) and never-smokers (group-2) with chronic periodontitis were included. Treatment wise, these individuals were divided into two subgroups as follows: (a) SRP alone and (b) SRP with adjunct aPDT. Periodontal parameters (plaque index [PI], bleeding on probing [BOP], clinical attachment loss [CAL] and probing pocket depth ≥4mm [PD] were measured at baseline and at 1 month and 3 months' follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported habitual cigarette-smokers.
* Self-reported never-smokers.
* Patients with chronic periodontitis (presence of at least 30% sites with ≥ 3 mm of CAL and PD ≥ 3 mm.

Exclusion Criteria:

* Patients with systemic diseases such as acquired immune deficiency syndrome/HIV and diabetes mellitus.
* Habitual smokeless tobacco product and alcohol users.
* Third molars and fractured teeth with embedded root remnants and edentulous individuals.
* Patients with misaligned teeth.
* Patients that reported to have used antibiotics, non-steroidal anti-inflammatory drugs and/or steroids within the past 90 days.

Ages: 42 Years to 52 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2017-07-02 (Actual); Study Completion 2017-09-16 (Actual)

PRIMARY OUTCOMES:
Probing depth | 3 months
  Probing depth will be measured as the distance from the gingival margin to the location of the tip of the probe to the nearest millimeter. Pocket depth assessment was carried out at 6 sites per tooth for all teeth (disto-buccal, mid-buccal, mesio-buccal, mesio-lingual, mid-lingual and disto-lingual)
Clinical attachment level gain | 3 months
  Clinical attachment level gain will be calculated for each site as the sum of probing depth and gingival recession. The CAL was recorded at 6 sites per tooth for all teeth (disto-buccal, mid-buccal, mesio-buccal, mesio-lingual, mid-lingual and disto-lingual) except third molars.

SECONDARY OUTCOMES:
Plaque index | 3 months
  Plaque index will be detected visually by running the probe at 4 sites per tooth (mesio-buccal, disto-buccal, mid-buccal and palatal/lingual) for absence or presence of plaque, based on dichotomous scoring system. The scores ranged as follows; 0 - No visible plaque
  1 - Visible plaque
Bleeding on probing | 3 months
  Bleeding on probing will be recorded at 4 sites per tooth (mesio-buccal, disto-buccal, mid-buccal, and palatal/lingual) for absence or presence of bleeding, based on dichotomous scoring system. The scores ranged as follows; 0 - No visible bleeding
  1 - Visible bleeding

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcome measures will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data is available